CLINICAL TRIAL: NCT01281943
Title: Phase II Study of Pegylated Liposomal Doxorubicin (Doxil®) and Temsirolimus (Torisel®) in Patients With Advanced Hepatocellular Cancer
Brief Title: Study of Pegylated Liposomal Doxorubicin and Temsirolimus in Patients With Advanced Hepatocellular Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Doxil Shortage
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201104170
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — temsirolimus; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus and Pegylated Liposomal Doxorubicin (Experimental): Temsirolimus 25mg andPegylated liposomal doxorubicin 25mg/m2
  Interventions: Drug: Temsirolimus 25mg and Pegylated liposomal doxorubicin 25mg/m2

INTERVENTIONS:
Drug: Temsirolimus 25mg and Pegylated liposomal doxorubicin 25mg/m2 — Temsirolimus 25mg IV on days 1, 8, 15 and 22 of each 28 day cycle
  Pegylated liposomal doxorubicin 25mg/m2 IV on day 1 of each 28 day cycle
  Other Names: (Torisel®); (Doxil®)

SUMMARY:
This Phase II study will use the MTD from a previous Phase I study at the recommended dose for the combination regimen from the Phase I trial, Doxil 25mg/m2 IV Q 4 weeks and temsirolimus 25mg IV Q week.

DETAILED DESCRIPTION:
This proposal aims to capitalize on the consensus recommendations of the NCI panel, the known antitumor activity of doxorubicin in HCC, and the as yet unpublished results of a recently completed Phase I clinical trial (WU HRPO# 07-0447, NCT00703170) combining pegylated liposomal doxorubicin (Doxil®) and temsirolimus (Torisel®) in patients with advanced solid tumors. In this Phase I study, twenty-two patients were enrolled and treated. The MTD and recommended Phase II dose for the combination regimen from this trial is is Doxil 25mg/m2 IV Q 4 weeks and temsirolimus 25mg IV Q week. During the conduct of this study two patients experienced confirmed partial responses (PR). One patient had heavily pretreated metastatic breast cancer and remained on the study for 6 months. The second patient with a PR had HCC that was previously treated with sorafenib. She remained on the study regimen for 14 months and tolerated this treatment well. Based on the tolerability of the drug combination and the observed anti-tumor activity in HCC, the current Phase II study in HCC is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Diagnosis: Patients must have a histologically or cytologically proven hepatocellular cancer (HCC) that is not amenable to treatment via resection or liver transplantation. In the absence of a tissue diagnosis, nodules on CT with a characteristic appearance of HCC plus Alpha Fetoprotein (AFP) > 400ng/ml will be considered diagnostic of HCC.
* Measurable Disease: Patients must have measurable disease.

Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques (PET, CT, MRI, x-ray) or as ≥10 mm with spiral CT scan. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters).

A positive bone scan, osteoblastic metastases, and pleural or peritoneal effusions are not considered measurable. Patients with only these lesions are not eligible for entry to the study.

* Prior Therapy: Patients may or may not have received prior systemic therapy in the metastatic setting. No prior treatment with an mTOR inhibitor or with doxorubicin is permitted. Participants must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. No chemotherapy or radiotherapy may be given within 4 weeks prior to the start of protocol treatment.
* Age: Patients must be ≥18 years old. Because no dosing or toxicity data are currently available on the use of temsirolimus in combination with pegylated liposomal doxorubicin in patients <18 years of age, children are excluded from this study.
* Performance Status: ECOG 0-2 at study entry.
* Life Expectancy: Patients must have a life expectancy of greater than 12 weeks.

Required Laboratory Values:

* absolute neutrophil count ≥1,500/mm3
* platelets ≥100,000/mm3
* hemoglobin ≥9.0 g/dL
* total bilirubin ≤1.5 x ULN
* AST(SGOT)/ALT(SGPT) ≤1.5 x ULN (≤2.5 x ULN for patients with liver metastases)
* alkaline phosphatase ≤2.5 x ULN
* creatinine ≤1.5 x ULN OR
* creatinine clearance ≥60 mL/min/1.732 for patients with creatinine levels above 2.0 mg/dl
* serum cholesterol ≤350 mg/dL /9.0 mmol/L (fasting)
* triglycerides ≤400 mg/dL (fasting)*
* albumin ≥3.0 mg/dL

  * Patients with triglyceride levels >400 mg/dL can be started on lipid lowering agents and reevaluated within 1 week. If levels go to ≤400 mg/dL, they can be considered for the trial and continue the lipid lowering agents.
  * Child-Pugh (CP) A or B liver dysfunction are eligible unless the bilirubin is >1.5 x ULN. If non-contraindicated, hepatic impairment (bilirubin >1-1.5 x ULN or AST >ULN but bilirubin ≤ULN) is present patients can be treated at a lower dose (15 mg/week) of temsirolimus.
* Concomitant Medications: Temsirolimus is primarily metabolized by CYP3A4. Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels. A partial list of agents which interact with cytochrome P450 (CYP3A) is found in Appendix B. Use of agents that potently inhibit CYP3A (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited. Temsirolimus can inhibit CYP2D6, and may decrease metabolism (and increase drug levels) of drugs that are substrates for CYP2D6, such as codeine. The appropriateness of use of such agents is left to physician discretion. A list of drugs that may have potential interactions with CYP2D6 is found in Appendix A. If there is any doubt about eligibility based on concomitant medication, the Principal Investigator should be contacted. All concomitant medications must be recorded.
* Known Allergies: Patients with known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin) are not eligible for this trial.
* Cardiac Function: Patients must have a normal left ventricular ejection fraction (LVEF ≥50%) by MUGA scan.
* Sexually Active Patients: For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential. Pregnant and nursing women are not eligible.
* HIV-Positive Patients: Patients receiving anti-retroviral therapy (HAART) for HIV infection are excluded from the study because of possible pharmacokinetic interactions. Appropriate studies will be undertaken in patients receiving HAART therapy, when indicated.
* Neurologic Status: Patients must not have active CNS disease.
* Recovery from Intercurrent Illness: Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Informed Consent: Patients must have signed a Washington University Human Research Protection Office (HRPO) approved informed consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
* Inclusion of Women and Minorities: Entry to this study is open to both men and women and to all racial and ethnic subgroups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 15 months
  To determine whether the progression free survival (PFS) rate in patients with advanced HCC using this combination regimen of pegylated liposomal doxorubicin and temsirolimus exceeds 5 months in the majority of treated patients, justifying the further development of this therapeutic regimen in this patient population.

SECONDARY OUTCOMES:
Toxicity and tolerability for this combination regimen | 3 months
  To further characterize the toxicity profile and tolerability for this combination regimen
Disease control rate, objective response rate, and overall survival. | 15 months
  To determine the disease control rate (DCR), objective response rate (ORR), and overall survival (OS) of this combination regimen
mTOR inhibition | 3 days
  To determine whether S6 kinase is inhibited in peripheral blood mononuclear cells (PBMCs) as an indication of adequate mTOR inhibitor exposure.
Pharmacogenomics | 1 day
  To measure Poly(ADP-ribose) polymerase-1 (PARP-1) activity in PBMCs from the patients as an indication of adequate doxorubicin exposure54.
Polymoprhism assessment | 1 day
  To assess whether common polymorphisms in ABCB1 and CYP2B6 are associated with any changes in treatment response or survival55.

CONTACTS AND LOCATIONS:
Overall Officials: A. Craig Lockhart, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu